CLINICAL TRIAL: NCT02896933
Title: Electrophysiological Study of Spatiotemporal Gait Parameters in Patients in Early Stage of Multiple Sclerosis
Acronym: MARCHE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RDZ_2014_17
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- patients with multiple sclerosis: recruited in a former study
- healthy control subjects

SUMMARY:
35 patients with multiple sclerosis have been enrolled in a previous study to record and analyze gait parameters.

This study aims to enroll gender and and matched healthy subjects for a control group, to compare patients' gait parameters with healthy subjects'.

ELIGIBILITY:
Inclusion Criteria:

* subjects without any gait trouble
* age ≥ 18 and < 55 years old
* gender and age (+/- 5 years) matched

Exclusion Criteria:

* pathology with potential gait impairment
* pregnant or breast feeding patient
* patient under legal protection
* no health insurance coverage
* absence of written informed consent

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 35 patients with multiple sclerosis progressing for less than 5 years, age 18 to 54 years old, and handicap score (EDSS) < 2 in all the subscores concerning gait, have been enrolled in a previous observational study recording and analyzing gait parameters.
  This study aims to enroll gender and aed matched healthy subjects for a control group, to compare patients' gait parameters with healthy subjects'.
  The 35 patients have given their consent for this new data analysis.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Variation coefficient of gait cadence | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël DEPAZ, MD, Principal Investigator — Fondation OPH A de Rothschild